CLINICAL TRIAL: NCT05462353
Title: A Phase II, Double-Blind, Randomized, Multicenter, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Efficacy of ASC41 in Subjects With Nonalcoholic Steatohepatitis (NASH)
Brief Title: Study to Evaluate the Safety, Tolerability, and Efficacy of ASC41 Tablets in Adult Patients With NASH
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gannex Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASC41-202
Record Dates: First submitted 2022-07-07; First posted 2022-07-18 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-10

CONDITIONS: Non-alcoholic Fatty Liver Disease; Non-alcoholic Steatohepatitis
Keywords: Non-alcoholic Fatty Liver Disease; NASH; ASC41; Phase II; THR-β
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 Low Dose (Experimental): 1 tablet of ASC41 (2 mg) for 52 weeks
  Interventions: Drug: 2mg of ASC41; Drug: Placebo
- Cohort 2 High Dose (Experimental): 2 tablet of ASC41 (4 mg) for 52 weeks
  Interventions: Drug: 4mg of ASC41 (2 tablets of 2 mg ASC41)
- Placebo tablet (Placebo Comparator): Placebo tablet for 52 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 2mg of ASC41 — ASC41 tablet administered orally once daily.
  Arms: Cohort 1 Low Dose
Drug: 4mg of ASC41 (2 tablets of 2 mg ASC41) — ASC41 tablets administered orally once daily.
  Arms: Cohort 2 High Dose
Drug: Placebo — Placebo tablets administered orally once daily.
  Arms: Cohort 1 Low Dose; Placebo tablet

SUMMARY:
This is a Phase 2, Double-Blind, Randomized, Multicenter, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Efficacy of ASC41 in Adults with Nonalcoholic Steatohepatitis (NASH).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 80 years old at screening.
* Presence of ≥ 7.5% steatosis on screening MRI-PDFF read centrally by a radiologist and performed either during the screening period or within 6 months prior to the first visit.
* HbA1c ≤ 9.5%.
* Normal or minimally abnormal renal function as defined by estimated glomerular filtration rate (eGFR) ≥ 50 mL/min/1.73 m^2

Exclusion Criteria:

* Presence or history of cirrhosis or evidence of decompensated liver disease (e.g., ascites, variceal bleeding) or hepatocellular carcinoma.
* History or presence of other concomitant liver disease as assessed by the investigator or determined by laboratory findings.
* Uncontrolled Type 2 diabetes mellitus (T2DM) defined as HbA1c of > 9.5% within 60 days prior to enrollment.
* Change in anti-diabetic therapy within 6 months prior to qualifying liver biopsy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2025-05-10 (Estimated); Study Completion 2025-06-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of ASC41 compared with placebo in noncirrhotic subjects with NASH by a histological change. | Baseline and Week 52
  A histological change in NAFLD (nonalcoholic fatty liver disease) Activity Score (NAS) ≥ 2 points that results from reduction of necroinflammation (inflammation or ballooning) without worsening fibrosis. (The NAFLD Activity Score including steatosis, inflammation and ballooning. The maximum score of steatosis was 3 and the minimum score was 0, the maximum score of inflammation was 3 and the minimum score was 0, and the maximum score of ballooning was 2 and the minimum score was 0. The higher scores mean a worse outcome. ）

SECONDARY OUTCOMES:
The incidence, type and severity of AEs/SAEs were assessed by CTCAE v5.0 to assess the safety and tolerability of ASC41 compared to placebo | 24 and 52 weeks
Change from baseline in hepatic fat fraction assessed by MRI-PDFF | 24 and 52 weeks
To evaluate the effect of ASC41 compared with placebo on serum lipids (cholesterol, HDL-C, LDL-C, triglycerides, Lp(a), VLDL) | 12, 24 and 52 weeks
Plasma pharmacokinetics - Peak Plasma Concentration (Cmax) | 1 and 15 Days
  Measured after administration
Plasma pharmacokinetics - Area under the plasma drug concentration versus time curve( AUC0-t_, AUC0-∞) | 1 and 15 Days
Plasma pharmacokinetics - The amount of time that a drug is present at the maximum concentration in serum(Tmax) | 1 and 15 Days

CONTACTS AND LOCATIONS:
Locations (1):
- The affiliated Hospital of Hangzhou Normal University, Hangzhou, Zhejiang, China